CLINICAL TRIAL: NCT05377554
Title: ALM-488 for Intra-Operative Visualization of Nerves in Head and Neck Surgery
Brief Title: Bevonescein for Intra-Operative Nerve Visualization in Head and Neck Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alume Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALM-488-002
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Surgery
Keywords: head and neck surgery; malignancy; thyroidectomy; parotidectomy; neck dissection; fluorescence; nerve; ALM-488; intra-operative; real-time
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This protocol describes prospective, open-label, blinded, randomized controlled, multicenter pivotal studies.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ALM-488-002a WLR only (Experimental): Patients with a preoperative diagnosis of malignancy will be assigned to study ALM-488-002a. All patients will receive ALM-488 infusion. Intraoperative nerve visualization will be performed using WLR only.
  Interventions: Drug: Bevonescein; Other: Intra-operative Visualization using White Light Reflectance (WLR)
- ALM-488-002a WLR with FL Overlay (Experimental): Patients with a preoperative diagnosis of malignancy will be assigned to study ALM-488-002a. All patients will receive ALM-488 infusion. Intraoperative nerve visualization will be performed using WLR with FL Overlay.
  Interventions: Drug: Bevonescein; Other: Intraoperative Visualization using White Light Reflectance (WLR) with Fluorescence (FL) Overlay
- ALM-488-002b WLR only (Experimental): Patients without a preoperative diagnosis of malignancy will be assigned to study ALM-488-002b. All patients will receive ALM-488 infusion. Intraoperative nerve visualization will be performed using WLR only.
  Interventions: Drug: Bevonescein; Other: Intra-operative Visualization using White Light Reflectance (WLR)
- ALM-488-002b WLR with FL Overlay (Experimental): Patients without a preoperative diagnosis of malignancy will be assigned to study ALM-488-002b. All patients will receive ALM-488 infusion. Intraoperative nerve visualization will be performed using WLR with FL Overlay.
  Interventions: Drug: Bevonescein; Other: Intraoperative Visualization using White Light Reflectance (WLR) with Fluorescence (FL) Overlay

INTERVENTIONS:
Drug: Bevonescein — Bevonescein will be infused during the pre-operative period.
  Other Names: ALM-488
Other: Intraoperative Visualization using White Light Reflectance (WLR) with Fluorescence (FL) Overlay — Intra-operative real time nerve visualization will be undertaken using WLR with FL Overlay.
  Arms: ALM-488-002a WLR with FL Overlay; ALM-488-002b WLR with FL Overlay
Other: Intra-operative Visualization using White Light Reflectance (WLR) — Intra-operative real time nerve visualization will be undertaken using WLR.
  Arms: ALM-488-002a WLR only; ALM-488-002b WLR only

SUMMARY:
This protocol describes prospective, open-label, blinded, randomized controlled, multicenter pivotal studies to evaluate ALM-488.

DETAILED DESCRIPTION:
This protocol describes prospective, open-label, blinded, randomized controlled, multicenter pivotal studies to evaluate ALM-488, a visualization adjunct for the real-time enhanced structural delineation of major nerves, in patients undergoing surgery of the Head and Neck.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a minimum of 16 years of age.
2. Must be planning to undergo surgery in the Head and Neck.
3. The study participant's primary surgical treatment is parotidectomy or thyroidectomy (unilateral or bilateral) or cervical neck dissection.
4. Willing and able to provide written assent as required and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
5. Willing and able to comply with all study procedures.
6. Sexually active patients must be willing to use an acceptable method of contraception (e.g., double barrier method) while participating in the study and for 30 days after receiving the last dose of ALM-488.
7. Females of childbearing potential must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had bilateral tubal ligation at least 1 year prior to screening, or who have had total hysterectomy.

Exclusion Criteria:

1. The patient has a history of prior radiation or surgery to the intended surgical site.
2. The patient has abnormal cardiac rhythm not controlled with medication.
3. The patient has moderate to severe renal impairment as indicated by a glomerular filtration rate (GFR) < 60 mL/min.
4. The patient has decreased hepatic function defined as aspartate aminotransferase (AST)/serum glutamic/oxaloacetic transaminase (SGOT) and alanine transaminase (ALT)/serum glutamic-pyruvic transaminase (SGPT) that is higher than 20% of the institution's normal laboratory limits, and/or the patient has elevated total bilirubin that is higher than 20% of the institution's normal laboratory limits.
5. The patient has unresolved acute toxicity from prior anti-cancer therapy grade 2 or higher, as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Alopecia, neuropathy ≤ Grade 2, as well as other non- acute and stable anti-cancer therapy toxicities are acceptable.
6. The patient has a history of fluorescein allergy.
7. The patient has a history of drug-related anaphylactic or severe allergic reactions.
8. Presence or history of any hypersensitivity to ALM-488 or its excipients that, in the judgment of the investigator, places the patient at increased risk for adverse effects.
9. Presence of a concurrent disease or condition that may interfere with study participation including recent (within 6 months of screening) NYHA Class III or IV heart failure, myocardial infarction (MI) or cerebrovascular accident (CVA).
10. Presence or history of any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.
11. Pregnant or breastfeeding at screening or planning to become pregnant (self or partner) at any time during the study.
12. Use of any Investigational Product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Contrast Enhancement | During surgery
  Nerve Contrast Enhancement will be compared between WLR and WLR with FL Overlay Using the Visualization Scoring System.
Length Measurement | During Surgery
  Nerve Length Measurement will be compared between WLR and WLR with FL Overlay Using a Metric Ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Orosco, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of California San Diego, La Jolla, California, United States